CLINICAL TRIAL: NCT01740401
Title: Phase II Study of CTLA-4 Blockade and Low Dose Cyclophosphamide in Patients With Advanced Malignant Melanoma
Brief Title: CTLA-4 Blockade and Low Dose Cyclophosphamide in Patients With Advanced Malignant Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary Endpoint not met
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Nina Bhardwaj, Director, Tumor Vaccine Program, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-0677; 114660 (Other: CA184-061)
Record Dates: First submitted 2012-11-29; First posted 2012-12-04 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-10

CONDITIONS: Melanoma
Keywords: Melanoma; Advanced Malignant Melanoma; Anti CTLA4 Blockade; Progression Free Survival; Interventional Therapy; Phase II Clinical Trial; Immunotherapy; T Cell Activation
MeSH Terms: conditions — Melanoma | interventions — Cyclophosphamide; Ipilimumab; CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide, Ipilimumab (Experimental): Treatment:
  Cyclophosphamide 300 mg/m2 po - Day 1 of Weeks 1, 4, 7, and 10, for a total of 4 doses; (premedication prior to each dose of Cyclophosphamide 8mg Zofran po, then prn)
  Ipilimumab 10 mg/kg iv - Day 3 of Weeks 1, 4, 7, and 10 for a total of 4 doses Maintenance treatment will be given on Weeks 24, 36, and 48 Ipilimumab 10 mg/kg iv
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — This study consists of a Treatment Period, D1 Zofran 8mg pre-Cyclophosphamide 300mg/mg2 po and D3 Ipilimumab 10mg/kg iv wks 1,4,7 and 10; Tumor assessment at week 12; Follow-Up period weeks 13,16,and 20 with no treatment; Maintenance Period, D1 10mg/kg iv wks 24,36,48 and 60. Week 40=end of treatment; week 60=end of study
  Other Names: Ipilimumab (BMS-734016, MDX010, MDX-CTLA4); Cytoxin

SUMMARY:
The purpose of this study is to see whether the combination of low-dose Cyclophosphamide and Anti-CTLA4 (Ipilimumab) will stop tumor growth in patients with advanced skin cancer. The investigators expect to see an increase in response rate of the combination over Anti-CTLA-4 alone and estimate a response rate of approximately 20 % in the proposed population.

DETAILED DESCRIPTION:
The transient removal of CTLA-4-mediated inhibition (CTLA-4 blockade) can induce effective anti-tumor immunity. Efficacy of CTLA-4 blockade as a single agent has been shown in melanoma 53. It has been hypothesized that anti-CTLA-4 antibody might deplete Treg cells 54, inducing autoimmunity. However, patients receiving Ipilimumab have not shown a decrease in Treg number or function in peripheral blood 55.

This trial will answer the question if the combination of Anti-CTLA 4 (following a well established regimen of Ipilimumab) and Cyclophosphamide (given at immunomodulatory doses) will result in antitumor activity in patients with metastatic melanoma due to synergistic immunomodulating effects by overcoming tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Men & women, ages ≥18
2. Willing/able to give written informed consent.
3. Histologic diagnosis of unresectable AJCC Stage III/IV malignant melanoma
4. At least 2wks must have elapsed since last chemotherapy, immunotherapy, hormonal therapy, radiotherapy or major surgery & beginning of protocol therapy. At least 6wks for nitrosoureas, mitomycin C, & liposomal doxorubicin
5. Toxicity related to prior therapy must either have returned to ≤ grade 1 or baseline.
6. Two punch tumor biopsy at Screening and Wk12 (4mm diameter) must be provided for immune analysis/staining if patients have accessible disease. Biopsies are optional during the Maintenance Period.Site of tumor biopsy s/n be only site of measurable disease. Minimum of 5 out of 1st 10 patients in stage I of the protocol must have biopsy accessible disease.
7. Patients must have measurable disease defined as @ least 1 lesion that can be accurately measured in @ least 1 dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
8. Required values for initial laboratory tests:

   1. WBC ≥ 2000/uL
   2. ANC ≥ 1000/uL
   3. Platelets ≥ 50 x 103/uL
   4. Hemoglobin ≥ 9.5 g/dL
   5. Creatinine ≤ 3.0 x ULN
   6. AST/ALT ≤ 2.5 x ULN for patients without liver metastasis, ≤ 5 x ULN for patients with liver metastasis
   7. Bilirubin ≤ 3.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
9. Life expectancy of at least 4mos
10. Patients w/stable, treated central nervous system (CNS) metastasis are eligible
11. ECOG Performance Status Score 0-1
12. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout study & for up to 26wks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized.

    WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not post-menopausal. Post-menopause is defined as:
    * Amenorrhea ≥ 12 consecutive months w/o another cause, or
    * For women with irregular menstrual periods and taking hormone replacement therapy (HRT), documented serum follicle-stimulating hormone (FSH) level ≥ 35 mIU/mL.
    * Women who are using oral contraceptives, other hormonal contraceptives (vaginal products/skin patches/implanted/injectable products), mechanical products such as an intrauterine device or barrier methods (diaphragm/condoms/ spermicides) to prevent pregnancy,are practicing abstinence or where their partner is sterile (eg vasectomy) should be considered to be of childbearing potential.
    * WOCBP must have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) w/in 72hrs before the start of ipilimumab.
13. Men of fathering potential must be using an adequate method of contraception to avoid conception throughout the study [and up to 26wks after last dose of investigational product] in a way that risk of pregnancy is minimized.

Exclusion Criteria:

1. Any other malignancy from which patient has been disease-free for less than 5yrs, with the exception of adequately treated & cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
2. Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (eg Guillain-Barre Syndrome and Myasthenia Gravis).
3. Any underlying medical or psychiatric condition, which in the opinion of investigator will make administration of ipilimumab hazardous or obscure interpretation of AEs, like a condition associated with frequent diarrhea.
4. Uncontrolled or significant cardiovascular disease
5. Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1mo before/after any dose of ipilimumab).
6. History of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist.
7. Concomitant therapy with any of following: IL 2, interferon, other non-study immunotherapy regimens; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (>60mg prednisone/day).
8. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg infectious) illness.
9. Women of childbearing potential (WOCBP), defined above who:

   1. are unwilling/unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 26wks after cessation of study drug, or
   2. have a positive pregnancy test at baseline, or
   3. are pregnant or breastfeeding.
10. Persons of reproductive potential who are unwilling to use an adequate method of contraception throughout treatment & for at least 26wks after ipilimumab is stopped.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Bhardwaj, MD,PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Clinical Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cyclophosphamide, Ipilimumab: Treatment:
  Cyclophosphamide 300 mg/m^2 po - Day 1 of Weeks 1, 4, 7, and 10, for a total of 4 doses; (premedication prior to each dose of Cyclophosphamide 8mg Zofran po, then prn)
  Ipilimumab 10 mg/kg iv - Day 3 of Weeks 1, 4, 7, and 10 for a total of 4 doses Maintenance treatment will be given on Weeks 24, 36, and 48 Ipilimumab 10 mg/kg iv
  Cyclophosphamide, Ipilimumab: This study consists of a Treatment Period, D1 Zofran 8mg pre-Cyclophosphamide 300mg/mg2 po and D3 Ipilimumab 10mg/kg iv wks 1,4,7 and 10; Tumor assessment at week 12; Follow-Up period weeks 13,16,and 20 with no treatment; Maintenance Period, D1 10mg/kg iv wks 24,36,48 and 60. Week 40=end of treatment; week 60=end of study
Period: Overall Study
Arm/Group | Cyclophosphamide, Ipilimumab
Started | 10
Completed | 0
Not Completed | 10
Not completed — Progression of disease | 6
Not completed — Adverse Event | 2
Not completed — Did not reach primary endpoint | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide, Ipilimumab
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 59 [36 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Malignant Melanoma (MM) site [Count of Participants; unit: Participants]
  Cutaneous MM | 7
  Ocular MM | 2
  Unknown Primary MM | 1

OUTCOME MEASURES:

1. Primary Outcome: The Anti-tumor Activity of the Combination of Low Dose Cyclophosphamide and CTLA-4 Blockade Using Objective Response Rate (ORR)
Description: Objective response rate (ORR) using mWHO RC. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, Ipilimumab
Number analyzed (Participants) | 10
Participants
  Stable disease | 4
  Progression of disease | 6

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is measured from date of entry to date of 1st documented evidence of recurrence, confirmation of PD, or death (whichever is 1st). T regulatory cells are measured on D1 (pre CTX) & D3 of each cycle.
Time Frame: Week 60
Population: Primary Endpoint not met, study terminated, data not collected
Arm/Group | Cyclophosphamide, Ipilimumab
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: Tumor-specific T Cell Responses Will be Measured in a Subset of Patients Who Have Biopsy Accessible Tumor and Have Tumor Biopsies Taken.
Description: One of the tumor punch biopsy will be put in formalin for paraffin-embedding. The other tumor punch biopsy will be processed to obtain lysates to be used as antigens for the T cell assays. Two tumor punch biopsies (4mm in diameter) will be obtained before and after therapy (baseline and week 12, and optional during weeks 24, 36, and 48) if patients have accessible tumors.
Time Frame: Week 48
Population: Primary Endpoint not met, study terminated, data not collected
Arm/Group | Cyclophosphamide, Ipilimumab
Number analyzed (Participants) | 0

4. Secondary Outcome: T Regulatory Cell Profile in Peripheral Blood
Description: Peripheral blood taken at baseline/various therapeutic time points/possibly maintenance cycles to evaluate T regulatory cells identified, serially monitored by polychromatic flow cytometry using FoxP3+/CD4+/CD127low/CD25hi markers.
Time Frame: Week 60
Population: Primary Endpoint not met, study terminated, data not collected
Arm/Group | Cyclophosphamide, Ipilimumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Cyclophosphamide, Ipilimumab: Treatment:
  Cyclophosphamide 300 mg/m^2 po - Day 1 of Weeks 1, 4, 7, and 10, for a total of 4 doses; (premedication prior to each dose of Cyclophosphamide 8mg Zofran po, then prn)
  Ipilimumab 10 mg/kg iv - Day 3 of Weeks 1, 4, 7, and 10 for a total of 4 doses Maintenance treatment will be given on Weeks 24, 36, and 48 Ipilimumab 10 mg/kg iv
  Cyclophosphamide, Ipilimumab: This study consists of a Treatment Period, D1 Zofran 8mg pre-Cyclophosphamide 300mg/mg2 po and D3 Ipilimuab 10mg/kg iv wks 1,4,7 and 10; Tumor assessment at week 12; Follow-Up period weeks 13,16,and 20 with no treatment; Maintenance Period, D1 10mg/kg iv wks 24,36,48 and 60. Week 40=end of treatment; week 60=end of study
Arm/Group | Cyclophosphamide, Ipilimumab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 4/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Ipilimumab (N=10)
Lipase elevation (Hepatobiliary disorders) | 1
Amylase elevation (Hepatobiliary disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Thromboembolic event (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide, Ipilimumab (N=10)
Anorexia (General disorders) | 1
Abdominal cramping (Gastrointestinal disorders) | 1
Depigmentation (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Lower back discomfort (Musculoskeletal and connective tissue disorders) | 1
Erythemia (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 4
Nausea (General disorders) | 3
Nasal congestion (General disorders) | 2
Pain (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes